CLINICAL TRIAL: NCT02185326
Title: Growth Hormone Co-treatment With the Microflare Stimulation Protocol in IVF/ICSI, Can it be a New Hope for Poor Responders?
Brief Title: Microflare Protocol in Poor Responders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Dina Mohamed Refaat Dakhly, Lecturer of obstetrics and gynecology, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WHE062013
Record Dates: First submitted 2014-07-01; First posted 2014-07-09 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Female Infertility Due to Diminished Ovarian Reserve
Keywords: Poor responders; Poor ovarian response; IVF/ICSI; Microflare protocol; Growth hormone; Oral contraceptive pills
MeSH Terms: interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Microflare and growth hormone (Experimental): the patients in this group were given oral contraceptive pills (OCPs) for 28 days, this was followed by 2 days free. Triptorelin (Decapeptyl Ferring Pharmaceuticals, Germany) 0.05 mg/day S.C. was then started daily followed by human menopausal gonadotropin IM daily (HMG 75 IU, Merional, IBSA) 3 days later. Growth hormone (Norditropin, Novo nordisk) was administrated on day 6 of HMG stimulation daily in a dose of 2.5 mg S.C. till the day of hCG administration.
  Interventions: Drug: Growth hormone (Norditropin, Novo nordisk)
- Microflare protocol alone (No Intervention): the patients in this group were given oral contraceptive pills (OCPs) for 28 days, this was followed by 2 days free. Triptorelin (Decapeptyl Ferring Pharmaceuticals, Germany) 0.05 mg/day S.C. was then started daily followed by human menopausal gonadotropin IM daily (HMG 75 IU, Merional, IBSA) 3 days later

INTERVENTIONS:
Drug: Growth hormone (Norditropin, Novo nordisk) — Growth hormone (Norditropin, Novo nordisk) was administrated on day 6 of HMG stimulation daily in a dose of 2.5 mg S.C. till the day of hCG administration.
  Other Names: Norditropin, Novo nordisk
  Arms: Microflare and growth hormone

SUMMARY:
The effect of use of the microflare down regulation protocol on the outcome of the IVF/ICSI cycles in poor responders

DETAILED DESCRIPTION:
The microflare as a method of down regulation protocol can be used to prepare the females suffering from poor ovarian reserve to undergo IVF/ICSI cycles. In this study we are trying to outline its effect on the clinical pregnancy rate as a main primary outcome, and to compare its use with the addition of growth hormone to the same protocol.

ELIGIBILITY:
Inclusion Criteria:

* females fulfilling the criteria of the ESHRE consensus 2011:

At least two of the following three features must be present:

(i) Advanced maternal age (≥40 years) or any other risk factor for POR; (ii) A previous POR (≤3 oocytes with a conventional stimulation protocol); (iii) An abnormal ovarian reserve test (i.e. AFC ,5-7 follicles or AMH ,0.5 -1.1 ng/ml).

Exclusion Criteria:

* women who suffer from any other cause of infertility other than poor ovarian reserve
* refusal of the patient to consent for using her data in the study.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rates | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Dakhly, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr el aini hospital, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Derived] Bayoumi YA, Dakhly DM, Bassiouny YA, Hashish NM. Addition of growth hormone to the microflare stimulation protocol among women with poor ovarian response. Int J Gynaecol Obstet. 2015 Dec;131(3):305-8. doi: 10.1016/j.ijgo.2015.05.034. Epub 2015 Aug 23. PMID 26381201